CLINICAL TRIAL: NCT01762579
Title: Not-celiac Wheat Sensitivity (NCWS) in Patients With Irritable Bowel Syndrome. Randomized Double-Blind Placebo-Controlled Trial (Wheat vs Placebo) for Bio-markers Identification of NCWS and Understanding Its Pathogenetic Mechanisms.
Brief Title: Bio-markers of Not-celiac Wheat Sensitivity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, MD, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: ACPM03
Record Dates: First submitted 2013-01-04; First posted 2013-01-07 (Estimated); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Not-celiac Wheat Sensitivity
Keywords: Not-celiac wheat sensitivity; Gluten; esophagogastroduodenoscopy; Rectoscopy
MeSH Terms: interventions — Flour; Xylose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- wheat flour (Active Comparator): wheat flour is administered blindly versus placebo for 15 days
  Interventions: Dietary Supplement: wheat flour; Dietary Supplement: Xylose
- Xylose (Placebo Comparator): placebo will be administered blindly versus wheat flour for 15 days
  Interventions: Dietary Supplement: wheat flour; Dietary Supplement: Xylose

INTERVENTIONS:
Dietary Supplement: wheat flour — wheat flour is administered three times per day for 15 days
Dietary Supplement: Xylose — Xylose will be administered three times per day for 15 days

SUMMARY:
The aim of the investigators' study is to evaluate biochemical, immunological and histological characteristics of patients affected with the so-called "gluten (or wheat) sensitivity" who suffers from irritable bowel syndrome (IBS)-like symptoms.

As it is not known what component of the cereals causes the symptoms in so called "gluten-sensitive" patients, the investigators prefer to speak of "not-celiac wheat sensitivity" (NCWS).

NCWS patients may be defined as ones, neither celiac or allergic to wheat, who develop symptoms following wheat consumption, that improved on wheat/gluten free diet (GFD). For our research, we will select adult patients, both genders, affected with suspected NCWS (i.e. with symptoms/signs which disappeared on GFD and worsen on a gluten containing diet, testing negative for celiac disease [anti-tissue transglutaminase antibodies, anti-tTG, and anti-endomysium antibodies, EMA, and with biopsy Marsh 0-1] and wheat allergy [serum specific IgE for wheat]). The patients will be recruited at the Department of Internal Medicine, 'Giovanni Paolo II' Hospital of Sciacca (Agrigento), and of Internal Medicine of the University of Palermo, from January 2012 to October 2013, for IBS-like symptoms.

At the time of the recruitment, the patients will be on GFD by at least one month and must be asymptomatic. A more restricted elimination diet (with the exclusion of cow's milk, egg and other foods) could be prescribed in patients who are suspected to suffer from multiple food hypersensitivity. The patients will be randomized to undergo a double-blind placebo-controlled study, assuming wheat flour or placebo, administered daily for 15 days. Before and after the challenge, the investigators will evaluate gastrointestinal (Gastrointestinal Symptom Rating Scale, GSRS) and the investigators will collect blood and fecal sampling and biopsies from endoscopic evaluation (both esophagogastroduodenoscopy and rectoscopy, with multiple biopsies), for the identification of possible markers (serological, biochemical, immunological, histological features, expression of cytokines and other constitutive mucosal proteins from peripheral blood mononuclear cells, mucosal lymphocytes and fecal biomarkers) that may be of help to diagnose the condition of NCWS and to understand its pathogenesis.

DETAILED DESCRIPTION:
Gluten is the most important protein component of some grains, notably wheat, rye, and barley, which are the basis for a variety of wheat-derived alimentary products consumed throughout the world (bread, pasta, pizza etc). However the "engineering" of gluten-containing grains created the conditions for human diseases related to gluten exposure. These forms of gluten intolerance represent a heterogeneous set of conditions, including celiac disease, wheat allergy and gluten sensitivity (GS), that, combined, seems to affect about 10% of the general population. The frequency of not-celiac GS is however still unknown, even though it is possible that this condition have been undiagnosed and under-diagnosed by the physicians for a long time. The immune responsiveness to wheat antigens represents a complex process, and its establishment and maintenance are not completely elucidated. The most frequent diseases caused by wheat ingestion are T cell-mediated disorders, i.e. celiac disease and IgE-mediated allergic reactions. However, besides celiac disease and wheat allergy, there are cases of gluten reactions in which neither autoimmune nor IgE-mediated allergic mechanisms are involved. These are generally defined as GS. Some subjects, who experience symptoms when eating gluten-containing products and show improvement when following a gluten-free diet (GFD), may have GS instead of celiac disease or wheat allergy. GS patients are unable to tolerate gluten and develop an adverse reaction when eating gluten, that, usually, and differently from celiac disease, does not lead to small intestinal damage. Gastrointestinal symptoms in GS patients may resemble those associated with celiac disease, but the overall clinical picture is generally less severe and is not accompanied by the occurrence of autoantibodies (i.e. anti-tTG or EMA) or autoimmune disease (i.e. Hashimoto's thyroiditis). Typically, the diagnosis is made by exclusion, and an elimination diet and an "open challenge" (i.e., the monitored reintroduction of gluten-containing foods) are most often used to evaluate whether health improves or worsen with the elimination or reintroduction of gluten in the diet, respectively. Gluten-sensitivity can cause both gastrointestinal and extra-intestinal symptoms; among the former, the most frequent are IBS-like symptoms including abdominal pain, bloating, diarrhea, constipation and alternate bowel habit. However, as it is not known what component of the cereals causes the symptoms in so called "gluten-sensitive" patients, we prefer to speak of "Not-celiac wheat sensitivity" (NCWS). Furthermore, in our experience, NCWS patients can suffer from multiple food hypersensitivity and need of a more restricted diet with the elimination of cow's milk, egg and other foods, in addition to wheat. For these reasons, before to undergo the gluten challenge, the patients will undergo an oligoantigenic diet.

This study has two major aims:

1. Evaluation of the effective dependence from the wheat of the IBS-like manifestations presented by subjects with suspected NCWS. The study will be done after a period of GFD, comparing two groups of suspected NCWS subjects: administering wheat flour or placebo (for 15 days).
2. Identification of possible markers (serological, biochemical, immunological, histological features, expression of cytokines and other constitutive mucosal proteins from peripheral blood mononuclear cells, mucosal lymphocytes and fecal biomarkers) that may be of help to diagnose the condition of NCWS. In particular, the investigators will search for markers of NCWS in the colon mucosa of the patients with IBS-like symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, both genders, with age between 18-65 years, with IBS-like symptoms, that improved on a gluten free diet and worsen on a gluten containing diet
* Patients testing negative for celiac disease ( anti-tTG and EMA negative, and with biopsy Marsh 0-1) and wheat allergy (serum specific igE for wheat negative)

Exclusion Criteria:

* Subjects diagnosed with celiac disease (positive anti-tTG and/or EMA, and positive histology, with Marsh 2 or above);
* Subjects diagnosed with wheat allergy (positive serum specific IgE for wheat)
* Subjects with Type 1 Diabetes
* Subjects with Inflammatory Bowel Diseases (Crohn's disease or ulcerative colitis)
* Subjects with Helicobacter pylori infection and other gastrointestinal infection
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Symptoms/signs evaluation | Change from baseline (i.e. before diagnosis of suspected NCWS, on free diet, and after diagnosis of suspected NCWS, on GFD) at 2 weeks
  Symptoms/signs evaluation, before and after the challenge: total score before and after 2 weeks of wheat (or placebo) ingestion

SECONDARY OUTCOMES:
Bio-Markers evaluation | Change from baseline (i.e. before diagnosis of suspected NCWS, on free diet, and after diagnosis of suspected NCWS, on GFD) at 2 weeks
  Bio-Markers to diagnose GS and understand its pathogenesis

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, PHD, MD, Principal Investigator — Internal Medicine, 'Giovanni Paolo II' Hospital of Sciacca (Agrigento) and University of Palermo, Palermo, Italy
Locations (2):
- Italy (2):
  - Internal Medicine, "Giovanni Paolo II" Hospital, Sciacca, Agrigento
  - Internal Medicine, University Hospital, Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seidita A, Giuliano A, Soresi M, Chiavetta M, Nardi E, Mogavero G, Giannone G, Carroccio A, Mansueto P. Fecal calprotectin levels in patients with non-celiac wheat sensitivity: a proof of concept. Intern Emerg Med. 2024 Aug;19(5):1255-1266. doi: 10.1007/s11739-024-03595-7. Epub 2024 Apr 12. PMID 38609737
- [Derived] Carroccio A, Giannone G, Mansueto P, Soresi M, La Blasca F, Fayer F, Iacobucci R, Porcasi R, Catalano T, Geraci G, Arini A, D'Alcamo A, Villanacci V, Florena AM. Duodenal and Rectal Mucosa Inflammation in Patients With Non-celiac Wheat Sensitivity. Clin Gastroenterol Hepatol. 2019 Mar;17(4):682-690.e3. doi: 10.1016/j.cgh.2018.08.043. Epub 2018 Aug 21. PMID 30138736